CLINICAL TRIAL: NCT07308106
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of SKB571 for Injection as Monotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With MET Abnormalities
Brief Title: A Phase II Clinical Study of SKB571 as Monotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With MET Abnormalities
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB571-Ⅱ-03
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non-small Lung Cancer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB571 monotherapy (Experimental)
  Interventions: Drug: SKB571 for injection

INTERVENTIONS:
Drug: SKB571 for injection — SKB571 for injection is administered every 3 weeks(Q3W) .

SUMMARY:
The aim of the study to evaluate the safety and efficacy of SKB571 for injection as monotherapy in patients with locally advanced or metastatic Non-Small Cell Lung Cancer with MET abnormalities. Eligible subjects will receive SKB571 monotherapy, until radiographic disease progression, intolerable toxicity, discontinuation of study treatment required by the subject, or other protocol-specified treatment discontinuation criteria, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤ 75 years at the time of signing the informed consent form (ICF).
2. Participants with histologically or cytologically confirmed NSCLC.
3. Locally advanced or metastatic NSCLC with MET Abnormalities that has progressed after standard therapy.
4. At least one measurable lesion as assessed by the investigator according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before the first dose.
6. Life expectancy ≥ 3 months as assessed by the investigator.
7. Adequate organ and bone marrow function.
8. Male and female participants must agree to use highly effective methods of contraception during the study treatment period.
9. Participants must voluntarily join this study, sign the ICF, and be able to comply with the visits and related procedures specified in the protocol.

Exclusion Criteria:

1. Participants with known active central nervous system (CNS) metastasis, and/or carcinomatous meningitis, brainstem metastasis, metastases to spinal cord, or spinal cord compression.
2. Participants with other malignant tumors within 3 years prior to the first dose.
3. Presence of any of the following cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
4. Presence of severe and/or uncontrolled concomitant diseases.
5. Participants with a history of interstitial lung disease (ILD) or a history of non-infectious pneumonitis.
6. Clinically severe lung damage due to complications of lung disorder.
7. Risk of esophagotracheal fistula or esophagopleural fistula, or tumor invasion or compression of surrounding vital organs and blood vessels.
8. Toxicity from prior anti-tumor therapy has not recovered to ≤ Grade 1.
9. Known active pulmonary tuberculosis.
10. Known history of allogeneic organ transplant or allogeneic hematopoietic stem cell transplant.
11. Active hepatitis B and hepatitis C.
12. Positive test for human immunodeficiency virus (HIV) or a medical history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
13. Known allergy or hypersensitivity to SKB571 or its excipients; or a history of severe allergy to other monoclonal antibodies.
14. Participants who have undergone major surgery within 4 weeks before the first dose or are expected to require major surgery during the study.
15. Serious infection within 4 weeks before the first dose.
16. Participants who have received systemic corticosteroid therapy with > 10 mg/day of prednisone or other immunosuppressive drugs within 2 weeks before the first dose of study treatment.
17. Participants who have received a live vaccine within 30 days before the first dose, or plan to receive a live vaccine during the study.
18. Pregnant or breastfeeding women.
19. Have local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors.
20. Any condition that, in the investigator's opinion, interferes with the evaluation of study treatment, participant safety, or interpretation of study results, or any other condition that the investigator deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
AE | Up to 24 months
  Incidence and severity of adverse events (AEs)
ORR | Up to 24 months
  Objective response rate (ORR) assessed by the investigator as per RECIST v1.1.

SECONDARY OUTCOMES:
DCR | Up to 24 months
  Disease control rate (DCR) (assessed by the investigators as per RECIST v1.1)
DOR | Up to 24 months
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
PFS | Up to 24 months
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
OS | Up to 24 months
  Time from start of treatment to death due to any reason.